CLINICAL TRIAL: NCT00768118
Title: A Pilot Study of Biomarker Alterations By Nutritional Agents
Brief Title: A Nutritional Supplement Capsule Containing Curcumin, Green Tea Extract, Polygonum Cuspidatum Extract, and Soybean Extract in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fazlul Sarkar, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000597010; P30CA022453 (NIH); WSU-2007-109; WSU-0211508MIE
Record Dates: First submitted 2008-10-04; First posted 2008-10-07 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Healthy, no Evidence of Disease
Keywords: healthy, no evidence of disease
MeSH Terms: interventions — Curcumin; Electrophoretic Mobility Shift Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Curcumin, Green Tea extract, Polygonum Cuspidatum & Soybean (Experimental): Total number of visits: 2, pre-intervention blood draw and urine sample collection, post-intervention blood draw and urine sample collection and interview Length of each visit: 15-30 minutes Total expected duration of participants' involvement: 15 days During the two-week intervention, volunteers will take two 1/2g capsules of the combination capsule, twice daily immediately after morning and evening meals.
  Interventions: Dietary Supplement: curcumin/green tea extract/Polygonum cuspidatum extract/soybean extract capsule; Genetic: electrophoretic mobility shift assay; Other: laboratory biomarker analysis

INTERVENTIONS:
Dietary Supplement: curcumin/green tea extract/Polygonum cuspidatum extract/soybean extract capsule
Genetic: electrophoretic mobility shift assay
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and urine from healthy participants receiving antioxidant nutritional supplements may help doctors identify changes in biomarkers related to oxidative stress.

PURPOSE: This clinical trial is studying how well a nutritional supplement capsule containing curcumin, green tea extract, Polygonum cuspidatum extract, and soybean extract works in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the effect of a specific combination nutritional capsule containing curcumin, green tea extract, Polygonum cuspidatum extract, and soybean extract on a specific biomarker of relevance to oxidative stress (NF-κB).
* To estimate the mean change in blood lymphocyte NF-κB level before and after 2 weeks of consumption of the nutritional agent under study.

OUTLINE: Participants receive oral curcumin/green tea extract/Polygonum cuspidatum extract/soybean extract capsule twice daily for 2 weeks. Participants are asked to keep a pill diary to track compliance.

Blood and urine samples are collected from participants at baseline and after completion of study. Lymphocytes and serum from the blood samples are isolated and analyzed for NF-κB biomarker levels. Urine samples are also tested for oxidative stress marker levels. Samples are analyzed using an electrophoretic mobility shift assay (EMSA).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Healthy volunteers who are employees of Karmanos Cancer Institute, Wayne State University, or Detroit Medical Center

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fazlul H. Sarkar, PhD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Biomarker Alterations by Nutritional Labels: Participants will donate a blood sample (pre & post intervention), two-3 tsp size tubes of blood will be collected in CPT tubes during each blood draw. Urine sample (pre & post intervention). During the 2-wk intervention period, the participant will be ingesting a nutritional supplement. Two capsules taken orally twice daily with meals, no other tests will be performed.
Period: Overall Study
Arm/Group | Biomarker Alterations by Nutritional Labels
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Biomarker Alterations by Nutritional Labels
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: The Magnitude of Change in Blood Lymphocyte NF-kB Level
Description: The target accrual goal is 15 subjects. It is hoped that of those 15, at least 10 will be intervention compliant, and provide both planned blood samples. NF-kB levels will be measured using a supershift assay, which tests the specificity and level of NF-kB in the sample by measuring the optical density of a scan. With 10 patients, the mean difference in blood lymphocyte NF-kB level could be estimated to within 0.44 standard 7 deviations, with 80% confidence. That is reasonable precision and confidence level for a small pilot study, and should provide sufficiently precise estimates for use in planning a subsequent study.
Time Frame: 15 days
Measure: Mean (90% Confidence Interval); unit: Optical Density unit
Arm/Group | Biomarker Alterations by Nutritional Labels
Number analyzed (Participants) | 9
Optical Density unit | -40.51 [-59.45 to -21.58]

ADVERSE EVENTS:
Arm/Group | Biomarker Alterations by Nutritional Labels
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
The study has small numbers, it was a proof-of-concept study only to demonstrate that agents taken orally can alter biomarkers, similar to the results obtained from in vitro studies, it was to open doors for future studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes